CLINICAL TRIAL: NCT05551819
Title: Acceptability of a Microbiome-directed Food for the Treatment of Children With Uncomplicated Acute Malnutrition in Niger
Brief Title: Acceptability of a Microbiome-directed Food in Young Children With Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Epicentre, Niger (Unknown); National Nutrition Direction, Niger (Unknown); Ministry of Public Health and Social Affairs, Niger (Unknown); Regional Direction of Public Health, Maradi (Unknown)
Responsible Party: Principal Investigator, Sheila Isanaka, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 823779-MDF Acceptability Niger
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feeding Order 1 (Experimental): MDF then RUTF/RUSF
  Interventions: Dietary Supplement: MDF then RUTF/RUSF
- Feeding Order 2 (Experimental): RUTF/RUSF then MDF
  Interventions: Dietary Supplement: RUTF/RUSF then MDF

INTERVENTIONS:
Dietary Supplement: MDF then RUTF/RUSF — Children randomized to feeding order 1: children will be provided MDF for the first two weeks then crossover to consume RUTF/RUSF for a second two weeks.
  Arms: Feeding Order 1
Dietary Supplement: RUTF/RUSF then MDF — Children randomized to feeding order 2: children will be provided RUTF/RUSF for the first two weeks then crossover to consume MDF for a second two weeks.
  Arms: Feeding Order 2

SUMMARY:
This study will compare the acceptability a microbiome-directed food (MDF) with standard formulations of therapeutic/supplementary foods for the treatment of acute malnutrition using a 2 x 2 crossover design.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted to assess the effectiveness of a microbiome-directed food (MDF) for treatment of uncomplicated acute malnutrition among children 6 to <24 months of age in Niger. MDF will be compared to standard ready-to-use therapeutic foods (RUTF) for children with severe acute malnutrition (SAM) and to standard ready-to-use supplementary foods (RUSF) for children with moderate acute malnutrition (MAM). The acceptability and utilization of MDF will be assessed in this preliminary acceptability study before the proposed effectiveness trial. The results of this preliminary acceptability study will be used to inform expectations of MDF use during the subsequent randomized effectiveness trial.

Children aged 6 to < 24 months will be eligible for enrollment in the acceptability trial on the day of their admission for treatment of uncomplicated severe or moderate acute malnutrition. Participants will be purposively selected to ensure balance by child age (6-11 vs 12 to < 24 months) and sex. Recruitment will occur continuously (e.g. without sampling on consecutive working days) among all eligible children at 2 study health centers until the target sample size is achieved.

After providing written informed consent, children will be randomized to 1 of 2 feeding orders (MDF vs RUTF/RUSF). Children will be randomized and provided with one product for the first two weeks then crossover to consume the second product for a second two weeks.

At each follow up visit, study nurses will ask caregivers rate their child's liking of the supplement on a 5-point Likert scale, as well as record child weight and any morbidity or adverse event since last visit before dispensing the next supply of food. Caregivers will also be asked to describe at-home utilization, including the food consumed by the child, current eating patterns in relation to other household foods (e.g. use at mealtimes, as a complete replacement, replacement of specific food items), sharing or selling practices in the home and willingness to use the supplement in the future.

ELIGIBILITY:
Inclusion Criteria:

* Are eligible for outpatient treatment of severe or moderate acute malnutrition according to the national protocol
* Are between 6 and <24 months of age
* Reside in the study catchment area and will remain there for at least 1 month
* Have no known allergy or contraindication to study product or standard treatment ingredients

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Acceptability of at-home ration | 2 weeks
  Consumption of 75% or more of the supplement provided during each 2-week period, where consumption is defined as total amount of food provided minus the total amount of food returned unused divided by the total amount of food provided.
Acceptability of test dose | 30 minutes
  Consumption of 75% or more of the test dose within 30 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Niger (2):
  - Guidan Roumji Health District, Guidan Roumji
  - Madarounfa Health District, Madarounfa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rattigan SM, Mbouombouo IN, Abdou Tahirou MA, Mostafa I, Saqeeb KN, Garba S, Guindo O, Ahmed T, Barratt MJ, Gordon JI, Sudfeld CR, Grais RF, Isanaka S. Acceptability of a Microbiome-Directed Food for the Management of Children with Uncomplicated Acute Malnutrition in Maradi, Niger: Two Randomized Crossover Trials. Curr Dev Nutr. 2025 Jun 9;9(7):107484. doi: 10.1016/j.cdnut.2025.107484. eCollection 2025 Jul. PMID 40672125